CLINICAL TRIAL: NCT05900479
Title: Multi-site, Longitudinal Trial Evaluating the Efficacy, Mechanisms, and Moderators of Service Dogs for Military Veterans With PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Maggie O'Haire, Associate Dean for Research, Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00002088; R01HD106413 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Stress Disorders, Post-Traumatic; Combat Stress Disorders; Animal-Human Bonding
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Human-Animal Bond

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD Service Dog (Experimental)
  Interventions: Other: PTSD Service Dog
- Usual Care (No Intervention)

INTERVENTIONS:
Other: PTSD Service Dog — According to the Americans with Disabilities Act (ADA), a service dog is a dog that is trained to perform specific tasks to mitigate a disability. For PTSD service dogs, examples include detecting and alerting to physical signs of distress to interrupt anxiety and panic attacks, waking up Veterans from nightmares, and retrieving medication. In addition to trained tasks, service dogs live with the Veterans to provide emotional value as a source of comfort and companionship. Under the ADA guidance, PTSD service dogs have pubic access and are legally allowed to accompany their person in public places such as grocery stores, workplaces, and schools. In the proposed study, service dogs will be sourced from three national service dog providers, including K9s For Warriors, Canine Companions, and America's VetDogs. All three providers have an established track record of training and providing service dogs for PTSD, as well as collaborating with the investigative team in research.
  Other Names: PTSD Assistance Dog; Psychiatric Service Dog
  Arms: PTSD Service Dog

SUMMARY:
Posttraumatic stress disorder (PTSD) among military Veterans is a critical public health concern. Veteran suicide rates exceed those of the general population, with the disorder creating a mental health challenge that is costly and debilitating. The majority of Veterans with PTSD also have comorbid mental health diagnoses, such as generalized anxiety disorder, substance abuse disorder, and major depression. The treatment of Veteran PTSD and comorbid disorders represents an important therapeutic and rehabilitation problem. The disorder is complex and difficult to treat, with high treatment dropout and nonresponse rates spurring some Veterans to seek complementary integrative health strategies. One promising complementary strategy is the provision of a trained service dog. Initial evidence across multiple research groups highlights service dogs as a promising complement to evidence-based practices that can offer short-term improvements. However, the long-term effectiveness, mechanisms of action, and moderators of efficacy remain largely unknown. Thus, the overarching objective of this proposal is to understand how, why, and for whom PTSD service dogs are most effective.

To address this objective, the present project will assess the longitudinal efficacy and dose-response curve of service dogs for Veteran PTSD symptomology and psychosocial functioning. The research design will consist of a two-arm, randomized clinical trial (RCT) with longitudinal assessments over a period of 15 months. Results are expected to elucidate the clinical impact of service dogs for military Veterans with PTSD, as well as the biobehavioral mechanisms of action and characteristics that moderate efficacy. These outcomes will support the long-term goal of accelerating complementary and integrative health interventions, through optimized and evidence-based service dog interventions. As such, this project will further advance the scientific understanding of human-animal interactions for psychosocial health.

ELIGIBILITY:
Inclusion Criteria:

* Applied for and approved to receive a psychiatric service dog from Canine Companions, K9s For Warriors, or America's VetDogs
* First service dog (not a successor service dog)
* Military service
* Honorable discharge or current honorable service
* Diagnosis of PTSD
* No conviction of any crimes against animals
* Able to follow the approved study timeline for randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
PTSD Severity and symptoms via self-report | 8 months
  Posttraumatic Stress Disorder Checklist for DSM-V (PCL-5, Range 0-80, Lower scores indicate a better outcome)

SECONDARY OUTCOMES:
PTSD Severity and symptoms via blinded clinician rating | 8 months
  Clinician-Administered PTSD Assessment for the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition DSM-V (CAPS-5-R, Range 0-80, Lower scores indicate a better outcome)
Depression | 8 months
  Patient Health Questionnaire (PHQ-9, Range 1-27, Lower scores indicate a better outcome)
Anxiety | 8 months
  Patient Reported Outcomes Measurement Information System (PROMIS) - Anxiety 8a (Raw Score Range 8-40, Lower scores indicate a better outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No